CLINICAL TRIAL: NCT00688363
Title: The Benefit of the Blood Glucose Self Monitoring and a Regular Three-monthly Hemoglobin A1c Profile in Patients With Type 2-diabetes and Conventional Insulin Therapy
Brief Title: Blood Glucose Self Monitoring and HbA1c Effects on Glucose Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsche Diabetes Gesellschaft (Other)
Collaborators: Bayer (Industry)
Responsible Party: Prof. Dr. M. Nauck, Kommission Klinische Studien der DDG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KKS 2003-Nauck-01
Record Dates: First submitted 2008-05-26; First posted 2008-06-02 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes control; glycated haemoglobin; blood-glucose-self-monitoring; type 2-diabetes; conventional insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): No blood-glucose self-control, no HbA1c
  Interventions: Procedure: no blood-glucose self-control
- 2 (Experimental): Blood-glucose self-control, no HbA1c
  Interventions: Procedure: weekly blood glucose profile
- 3 (Experimental): No blood-glucose self-control, HbA1c
  Interventions: Procedure: three-monthly haemoglobin A1c; Procedure: no blood-glucose self-control
- 4 (Experimental): Blood-glucose self-control, HbA1c
  Interventions: Procedure: weekly blood glucose profile; Procedure: three-monthly haemoglobin A1c

INTERVENTIONS:
Procedure: weekly blood glucose profile — once daily self-control of urinary-glucose
  Arms: 2; 4
Procedure: three-monthly haemoglobin A1c — once daily self-control of urinary-glucose
  Arms: 3; 4
Procedure: no blood-glucose self-control — once daily self-control of urinary-glucose
  Arms: 1; 3

SUMMARY:
The purpose of this randomized, prospective trial is to determine wether (a) a once weekly glucose profile (self monitoring) or (b) a three-monthly report of the actual glycated haemoglobin are effective interventions to improve HbA1c after one year in typ 2-diabetic patients on conventional insulin treatment.

DETAILED DESCRIPTION:
The design is an open, prospective, randomised, multicentre parallel group study. The total duration will be 5 years with patient recruitment over 4 years and an individual observation period of 1 year. 300 participants from 43 study centres, hospitals and private practices were recruited. The study will run for one year and aims to determine, whether there is an advantage with regard to HbA1c levels when (a) a regular three-monthly HbA1c or (b) a weekly 4-point glucose profile is taken and reported.

After screening, patients will be assigned at random to one of the following study arms:

1. no regular blood-glucose self-monitoring, no regular HbA1c
2. regular blood glucose self monitoring, no regular HbA1c
3. no regular blood glucose self monitoring, regular HbA1c
4. regular blood glucose self monitoring, regular HbA1c

The control for all participants is that urinary glucose should be monitored at least once a day, preferably in the late morning, as the highest increase in plasma glucose level occurs after breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Type 2-diabetes (ADA/WHO-Criteria)
* Conventional insulin therapy ( 1-3 daily injections of basal- and/or mixed insulin also in combination with oral agents.)
* Age:> 40 years
* BMI:> 20 kg/m²

Exclusion Criteria:

* Impaired liver function, defined as > 2 times upper limit of normal
* Impaired renal function defined liver enzymes as serum-creatinine > 1.3 mg/dl
* Gastro-intestinal diseases (disturbances, diagnoses)
* Inability to perform study-related activities according to the present protocol
* Pregnancy not certainly excluded
* Abuse of alcohol and/or other drugs
* Participation in other clinical trials during the past 3 month
* Threat to general state of health
* Intensified insulin therapy (at least 3 times rapid-acting insulin)
* Frequent blood glucose self monitoring during the past 3 months (more than one 4-point glucose profile per week or more than one blood glucose/ urinary glucose test per day )

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-02; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Haemoglobin A1c after one year | 1 year

SECONDARY OUTCOMES:
a representative blood glucose profile (self monitoring) during the week before the end of the trial | 1 year
body weight at the end of the trial | 1 year
serum, triglycerides and cholesterol (total HDL as well as LDL-cholesterol) at the end of the trial | 1 year
therapy-satisfaction (questionnaire) | 1 year
changes of the antidiabetic therapy | 1 year
number of hospitalization as a result of hypoglycaemic episodes | 1 year
the number of serious hypoglycaemic episodes (hypoglycaemic episodes when the patient needs help from other people) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof. Dr., Principal Investigator — Diabeteszentrum Bad Lauterberg
Locations (41):
- Germany (41):
  - Diabeteszentrum Bad Lauterberg, Bad Lauterberg im Harz, Lower Saxony
  - Koch, Peter, Bad Harzburg
  - Maxeiner, Stefan, Bad Kreuznach
  - Friedrichs, Michael, Bad Lauterberg im Harz
  - Jödicke, Carmen, Bad Lauterberg im Harz
  - Mulch-Wiemer, Christa, Bad Nauheim
  - Bellmann, Renate, Berlin
  - Schoch, Daniela, Berlin
  - Warmers, Ulrike, Bitburg
  - Leupold, Manfred, Borna
  - Kamke, Wolfram, Burg/Sreewald
  - Hildebrandt, Rüdiger, Clausthal-Zellerfeld
  - Lemmerhirt, Jürgen, Cuxhaven
  - Preuß, Uwe, Datteln
  - Weller, Ulrich, Dorsten
  - Fischer, Harald, Düren
  - Krege, Peter, Emsdetten
  - Gölz, Stefan, Esslingen am Neckar
  - Wollersen, Karin, Freiburg im Breisgau
  - Hendel, Andreas, Grassau
  - Pfeiffer, Martha, Gronau
  - Jäger, Michael, Höchst
  - Müller, Ulrich. A., Jena
  - Niemetz, Ingo, Kassel
  - Schmitz, Ulrike, Krefeld
  - Kourbanova, Zarema, Langenfeld
  - Willms, Gerhard, Leverkusen
  - Ley, Heinz-Georg, Marl
  - Grossmann, J., Mönchengladbach
  - Füchtenbusch, Martin, München
  - Fueting, Frank, Nassau
  - Behnke, Thomas, Neuwied
  - Böhme, Rainer, Nordhausen
  - Fels, Stefan, Oldenburg
  - Klein, Frank, Schenklengsfeld
  - Naumann, Rainer, Schöppenstedt
  - Rieth-Kunert, Anna, Stade
  - Nowack, Kirsten, Torgau
  - Schmidt-Reinwald, Astrid, Waldrach
  - Bödecker, A.-W., Wiehl
  - Oerter, Erika-Maria, Würzburg

REFERENCES:
- [Derived] Nauck MA, Haastert B, Trautner C, Muller UA, Nauck MA, Heinemann L; Clinical Trials Study Group of the German Association for the Study of Diabetes (Deutsche Diabetes-Gesellschaft). A randomised, controlled trial of self-monitoring of blood glucose in patients with type 2 diabetes receiving conventional insulin treatment. Diabetologia. 2014 May;57(5):868-77. doi: 10.1007/s00125-014-3168-1. Epub 2014 Jan 21. PMID 24445534